CLINICAL TRIAL: NCT04836364
Title: Prevalence of Endocrine Disorders Among Children Exposed to Lavender Essential Oil and Tea Tree Essential Oils
Brief Title: Skincare Products and Environmental Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 19-03-1700
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Gynecomastia; Endocrine System Diseases
Keywords: Prepubertal Gynecomastia; Essential Oils; Lavender; Tea Tree; Endocrine Disruption; Pediatric Environmental Health
MeSH Terms: conditions — Gynecomastia; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Cohort: Parents of children ages 2 to 15 years old will provide data using the APICHS.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention; observation only.

SUMMARY:
The purpose of this study is to explore the potential for an association between the development of prepubertal gynecomastia and history exposure to lavender essential oil, tea tree essential oil, and other essential oils.

DETAILED DESCRIPTION:
After being informed about the study and privacy, parents will give informed consent and complete the APICHS (Aromatic Plant Ingredient & Child Health Survey), a validated measurement tool for determining exposure to plant-based ingredients in pediatric personal care products.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child aged 2-15 living in the United States

Exclusion Criteria:

* none

Ages: 2 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Parents of children aged 2 to 15 years old who live in the United States will be recruited for this study. Emphasis is placed on obtaining a diverse sample which all states and territories, in addition to a racially and SES diverse sample.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lifetime prevalence of prepubertal gynecomastia | Baseline
  The number of participants who were exposed to lavender and tea tree essential oils and had ever experienced prepubertal gynecomastia
Lifetime prevalence of precocious puberty | Baseline
  The number of participants who were exposed to lavender and tea tree essential oils and experienced prepubertal gynecomastia
Endocrine Disruption - Comparison between exposed and unexposed | Baseline
  The difference in rates of endocrine disorders between children who were exposed to lavender or tea tree essential oil and those who were not. Exposure is measured using the Aromatic Plant Ingredient and Child Health Survey (APICHS), which measures total exposure, providing a continuous variable ranging from 0 to unlimited exposures, and a dichotomous yes/no exposure outcome variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No